CLINICAL TRIAL: NCT04702815
Title: Post-Stroke Visual Dependence and Early Intervention of Multisensory Balance Rehabilitation
Brief Title: Visual Dependence and Multisensory Balance Rehabilitation After Stroke
Status: Completed | Type: Observational
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Shu-Chun Lee, Principal Investigator, Taipei Medical University
Other Study IDs: N201912127
Record Dates: First submitted 2020-12-08; First posted 2021-01-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Stroke; Balance; Distorted; Gait, Unsteady
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cross-sectional study aims to investigate the prevalence of post-stroke visual dependence, and the effects of visual dependence on balance and gait. It also determines whether visual dependence could differentiate stroke patients with a history of falls from without.

DETAILED DESCRIPTION:
Stroke participants will be recruited to measure the level of visual dependence, muscle strength, neurological recovery, balance ability, vertigo symptom, gait pattern and activities of daily living. This will calculate the prevalence of post-stroke visual dependence, and investigate the negative impact of visual dependence on balance and walking functions. This also determines whether the value of visual dependence could differentiate stroke patients with a history of falls from without a history of falls.

ELIGIBILITY:
Inclusion Criteria:

* 1) first stroke with 20-80 years of age
* 2) the time since onset is more than 6 months
* 3) can walk independently at least 10 meters without any walking devices and orthosis
* 4) normal cognitive function with scoring more than 24 on the Mini Mental State Examination scale
* 5) can understand and follow commands
* 6) can give informed consent

Exclusion Criteria:

* 1) other neurological disorders which could affect balance assessment
* 2) cerebellar stroke
* 3) diagnosis with central or peripheral vestibular diseases.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic stroke patients with the first stroke will be recruited from the 3 departments of physical and rehabilitation medicine, regional hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Perceived visual dependence | Baseline
  Perceived visual dependence will be assessed using a computerized Rod and Disc Test (RDT). Participants will adjust a tilted rod to their subjective visual vertical with rotating visual background. The error (degrees) between subjective visual vertical and gravitational vertical will be measured and represented as the level of visual dependence. Higher error indicates higher level of perceived visual dependence.
Postural visual dependence | Baseline
  Postural sway will be measured using an accelerometer attached on the lower back when participants are looking at blank wall, eyes closed and looking at rotating visual background. Greater postural sway in conditions with eyes closed and rotating visual background corresponding to looking at blank wall represents the higher level of postural visual dependence.
A history of falls | Baseline
  Any falls in the past year (n). Fall is defined by the inadvertently coming to rest on the ground, floor or other lower level, excluding intentional change in position to rest in furniture, wall or other objects. More than once fall is identified as faller.

SECONDARY OUTCOMES:
Physical impairment of paretic leg and foot | Baseline
  Physical impairment of paretic leg and foot will be assessed by the Chedoke-McMaster Stroke Assessment (CMSA) with scoring on a 7-point scale (Stage 1 through 7, most impairment through to no impairment, respectively). The higher stage indicates the better neurological recovery.
Five Times Sit to Stand Test | Baseline
  The five Times Sit to Stand Test (5STS) evaluates functional lower extremity strength. Participants will be asked to sit to stand for 5 times as quickly as possible. The time to complete the task will be recorded. The shorter duration (s) represents the better muscle strength in lower limbs.
Berg Balance Scale | Baseline
  The Berg balance scale (BBS) is used to objectively determine a participant's ability to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. The total score is 56.
Timed Up and Go test | Baseline
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. The longer duration (s) to complete the task represents the poorer balance.
Modified Clinical Test of Sensory Integration and Balance | Baseline
  Modified Clinical Test of Sensory Integration and Balance (mCTSIB) is designed to assess how well an older adult is using sensory inputs when one or more sensory systems are compromised. Postural sway will be measured using an accelerometer attached on the lower back in 4 sensory conditions with visual and proprioceptive manipulation.
Falls Efficacy Scale - International | Baseline
  Falls Efficacy Scale- International (FES-I) assesses subjects' concerns about falling. It consists of 16 questions related to everyday activities and subjects are asked to rate whether they were "not at all" (a score of 1), "somewhat" (2), "fairly" (3) or "very" (4) concerned about falling when doing that particular activity. The sum scores ranged 16 - 64 with higher scores indicating a greater fear of falling.
Situational Vertigo Questionnaire | Baseline
  The Situational Vertigo Questionnaire (SVQ) is a 19-item questionnaire specifically aimed at identifying the presence of visual vertigo, a condition attributable to a defective vestibular compensation strategy, which is too dependent on the available visual information. Higher score represents more severe vertigo symptoms.
Gait pattern | Baseline
  Gait pattern will be evaluated using a Opal wireless system. Participants will be asked to walk in a 14-meter walkway. The first and final 2 meters are designed for acceleration and deceleration. The middle 10-meter will be analyzed only.
Barthel index | Baseline
  The Barthel Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored. The total score is 100 and higher score represents more independent in ADL.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chun Lee, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan